CLINICAL TRIAL: NCT00607906
Title: A Single-blinded, Randomized, Placebo-controlled, Staggered-parallel, Escalating Single Dose Study to Investigate the Safety, Tolerability, Pharmacokinetics and Pharmacodynamics of Orally Administered SB756050 in Healthy Volunteers and in Subjects With Type 2 Diabetes Mellitus
Brief Title: First-Time-in-Humans Study to Assess Safety, Pharmacokinetics & Pharmacodynamics of SB756050
Status: Completed | Phase: Phase 1 | Type: Interventional
Sponsor: GlaxoSmithKline (Industry)
Responsible Party: Sponsor
Allocation: Randomized | Model: Parallel | Purpose: Treatment
Other Study IDs: AXO110461
Record Dates: First submitted 2008-01-23; First posted 2008-02-06 (Estimated); Last update posted 2017-09-06 (Actual); Status verified 2017-09

CONDITIONS: Diabetes Mellitus, Type 2
Keywords: safety; pharmacodynamics; diabetes; pharmacokinetics
MeSH Terms: conditions — Diabetes Mellitus, Type 2; Diabetes Mellitus

STUDY DESIGN:
Oversight: Data Monitoring Committee: No

ARMS (5):
- Subjects receiving treatment in cohort A1 (Experimental): Eligible subjects will receive oral immediate release capsules of SB-756050 with doses of 5 milligrams, 15 milligrams, 50 milligrams, or 100 milligrams.
  Interventions: Drug: SB-756050 immediate release capsule; Drug: Placebo
- Subjects receiving treatment in cohort A2 (Experimental): Eligible subjects will receive oral immediate release capsules of SB-756050 with doses of 100 milligrams, 200 milligrams, 300 milligrams, or 400 milligrams.
  Interventions: Drug: SB-756050 immediate release capsule; Drug: Placebo
- Subjects receiving treatment in cohort A3 (Experimental): Eligible subjects will receive oral immediate release capsules of SB-756050 with a dose of 150 milligrams. Subjects will also receive oral modified release capsules of SB-756050 with doses of 150 milligrams, 300 milligrams, or 400 milligrams.
  Interventions: Drug: SB-756050 immediate release capsule; Drug: SB-756050 modified release capsule; Drug: Placebo
- Subjects receiving treatment in cohort A4 (Experimental): Eligible subjects will receive SB-756050 in this additional cohort.
  Interventions: Drug: SB-756050 immediate release capsule; Drug: Placebo
- Subjects receiving treatment in cohort B1 (Experimental): Eligible subjects will receive oral modified release capsules of SB-756050 with doses of 50 milligrams, 150 milligrams or 400 milligrams. Subjects will also receive immediate release oral capsules of SB-756050 with a dose of 150 milligrams.
  Interventions: Drug: SB-756050 immediate release capsule; Drug: SB-756050 modified release capsule; Drug: Placebo

INTERVENTIONS:
Drug: SB-756050 immediate release capsule — SB-756050 immediate release capsules will be size 0, white, opaque capsules with no identifying markings, containing white to off-white drug layered pellets. Each capsule will contain 5, 25 or 100 milligrams of SB-756050.
Drug: SB-756050 modified release capsule — SB-756050 modified release capsules will be size 0, white, opaque capsules with no identifying markings, containing white to off-white enteric coated drug layered pellets. Each capsule will contain either 25or 100 milligrams of SB-756050.
  Arms: Subjects receiving treatment in cohort A3; Subjects receiving treatment in cohort B1
Drug: Placebo — Subjects will also receive placebo capsules.

SUMMARY:
This study will use single escalating doses of SB756050 to assess safety, pharmacokinetics, and pharmacodynamics in healthy volunteers and in subjects with Type 2 Diabetes Mellitus.

ELIGIBILITY:
Inclusion Criteria:

Healthy Subjects

* Healthy male or female subject as determined by a responsible physician, based on a medical evaluation including history, physical examination, vitals signs, laboratory tests, and cardiac monitoring.
* Female subjects must be of non-childbearing potential including pre-menopausal women with documented (medical report verification) hysterectomy, tubal ligation, or postmenopausal defined as 12 months of spontaneous amenorrhea or 6 months of spontaneous amenorrhea with serum FSH levels > 40 mIU/ml or 6 weeks postsurgical bilateral oophorectomy with or without hysterectomy.
* 18 - 60 years of age, inclusive, at the time of signing and dating the informed consent.
* BMI (body mass index) within the range 20-30 kg/m2, inclusive.
* Capable of giving written informed consent, which includes compliance with the requirements and restrictions listed in the consent form.

Diabetic Subjects

* Male or female subjects, 18 - 60 years of age, inclusive, at the time of signing the informed consent
* Female subjects must be of non-childbearing potential including pre-menopausal women with documented (medical report verification) hysterectomy, tubal ligation, or double oophorectomy or postmenopausal defined as 12 months of spontaneous amenorrhea or 6 months of spontaneous amenorrhea with serum FSH levels > 40 mIU/ml or 6 weeks postsurgical bilateral oophorectomy with or without hysterectomy.
* Subjects should have no significant known medical conditions other than T2DM.
* BMI (body mass index) within the range 25-35 kg/m2, inclusive.
* T2DM diagnosed at least 3 months prior to Screening with

  * Fasting plasma glucose (FPG) level ≤ 220mg/dL at the Screening visit,
  * FPG level ≤ 250 mg/dL on Day -1 of Period 1
  * For subjects taking no antidiabetic medications: HbA1c between 7 and 10%, inclusive, at Screening visit
  * For subjects taking metformin or a sulfonylurea: HbA1c between 6.5 and 9.5%, inclusive, at Screening visit
* Subjects must be taking either no anti-diabetic medication, or metformin as monotherapy, or a sulfonylurea as monotherapy. (Subjects taking BOTH metformin and a sulfonylurea are not qualified for the trial). If taking metformin or a sulfonylurea, the dose must have been stable for at least 3 months prior to screening, and the subject must be willing to wash out from metformin or sulfonylureas from Day -7 prior to Period 1, through discharge from Period 4.
* Capable of giving written informed consent, which includes compliance with the requirements and restrictions listed in the consent form.

Exclusion Criteria:

* As a result of the medical interview, physical examination, or screening investigations, the Investigator considers the subject unfit for the study.
* Has any of the following laboratory abnormalities:

  * Positive pre-study Hepatitis B surface antigen, positive Hepatitis C, or HIV result.
  * History of uncorrected thyroid dysfunction or an abnormal thyroid function test assessed by TSH at Screening
  * A positive pre-study drug/urine screen. A minimum list of drugs that will be screened for include amphetamines, barbiturates, cocaine, opiates, cannabinoids and benzodiazepines.
  * A pre-study urine cotinine screen indicating use of tobacco/ nicotine containing products.
* Has a history of any gastrointestinal or hepatic conditions that could impact absorption of the investigational compound.
* Has QTc at Screening > 450 msec. Note that if the initial QTc value is prolonged, the ECG should be repeated two more times (with 5 minutes between ECG readings) and the average of the 3 QTc values used to determine eligibility.
* Has clinically significant rhythm abnormalities identified during 24-hour Screening Holter assessment.
* History of regular alcohol consumption averaging >7 drinks/week for women or >14 drinks/week for men. One drink is equivalent to 12 g alcohol (which equals 5 ounces (150 mL) of wine, 12 ounces (360 mL of beer or 1.5 ounces (45 mL) of 80 proof distilled spirits) within 6 months of screening.
* Smoked or used tobacco or nicotine-containing products within the previous 6 months.
* Has participated in a clinical trial and has received a drug or a new chemical entity within 30 days or 5 half-lives, or twice the duration of the biological effect of any drug (whichever is longer) prior to the first dose of current study medication.
* Exposure to more than four new chemical entities within 12 months prior to the first dosing day.
* Use of prescription or non-prescription drugs, including vitamins, herbal and dietary supplements (including St John's Wort) within 7 days or 5 half-lives (whichever is longer) prior to the first dose of study medication. Acetaminophen may be used as needed for adverse events; however, use should be restricted to 4 hours after dosing if possible with a preferred maximum dose of 2 grams in 24 hours.
* Unwilling to abstain from

  * Caffeine-or xanthine-containing products for 24 hours prior to dosing until the final post-dose assessment at each treatment level.
  * Use of illicit drugs
  * Alcohol for 24 hours prior to dosing until final post-dose assessment at each treatment level.
  * Consumption of red wine, Seville oranges, grapefruit or grapefruit juice from 7 days prior to the first dose of study medication until collection of the final pharmacokinetic and pharmacodynamic blood samples.
* History of sensitivity to any of the study medications, or components thereof or a history of drug or other allergy that, in the opinion of the physician responsible, contraindicates their participation. This includes sensitivity to heparin, if heparin will be used to maintain catheter patency.
* Where participation in the study would result in donation of blood in excess of 500 mL within a 56 day period.
* Subject is either an immediate family member of a participating investigator, study coordinator, employee of an investigator; or is a member of the staff conducting the study.

Healthy Subjects

* As a result of the medical interview, physical examination, or screening investigations, the Investigator considers the subject unfit for the study.
* Has any of the following laboratory abnormalities:

  * Positive pre-study Hepatitis B surface antigen, positive Hepatitis C, or HIV result.
  * History of uncorrected thyroid dysfunction or an abnormal thyroid function test assessed by TSH at Screening. (NOTE: subjects with hypothyroidism on a stable dose of thyroid replacement therapy for at least 3 months prior to Screening and who have a screening thyroid stimulating hormone (TSH) within the normal range may participate.)
  * ALT and/or AST > 2 times the upper limit of normal at screening or prior to the first dose.
  * Fasting triglycerides > 450mg/dL at screening or prior to the first dose.
  * Total Bilirubin > 1.5 times the upper limit of normal at screening or prior to the first dose
  * A positive pre-study drug/urine screen. A minimum list of drugs that will be screened for include amphetamines, barbiturates, cocaine, opiates, cannabinoids and benzodiazepines.
  * A pre-study urine cotinine screen indicating use of tobacco/ nicotine containing products.
* Significant renal disease or loss of a kidney
* Significant ECG abnormalities,
* Systolic pressure > 150 mmHg or <80 mmHg or diastolic blood pressure > 95 mmHg or <60 mmHg at screening. Blood pressure assessments may be repeated once if needed, allowing adequate time for subject to rest.
* Previous use of insulin as a treatment within 3 months of Screening, or for >2 weeks when used for acute illness in the last 12 months prior to Screening, or if used for more than 1 year when associated with GDM.
* Has a history of any of the following conditions:

  * Clinically significant symptoms of gastroparesis
  * Cholelithiasis or obstructive or inflammatory gallbladder disease within 3 months prior to Screening
  * Gastrointestinal disease that could affect fat or bile acid absorption, including inflammatory bowel disease, chronic diarrhea, Crohn's or malabsorption syndromes within the past year
  * Gastrointestinal surgery
  * Chronic or acute pancreatitis
* History of regular alcohol consumption averaging >7 drinks/week for women or >14 drinks/week for men. 1 drink is equivalent to (12 g alcohol) = 5 ounces (150 mL) of wine or 12 ounces (360 mL) of beer or 1.5 ounces (45 mL) of 80 proof distilled spirits) within 6 months of screening.
* Smoked or used tobacco or nicotine-containing products within the previous 6 months.
* Has participated in a clinical trial and has received a drug or a new chemical entity within 30 days or 5 half-lives, or twice the duration of the biological effect of any drug (whichever is longer) prior to the first dose of current study medication.
* Exposure to more than four new chemical entities within 12 months prior to the first dosing day.
* Is taking prohibited medications:

  * Acetaminophen may be used as needed for adverse events; however, use should be restricted to 4 hours after dosing if possible with a preferred maximum dose of 2 grams in 24 hours.
  * The use of anti-diabetic agents other than metformin or sulfonylureas is reason for exclusion and subjects will not be allowed to wash off of unapproved anti-diabetic medications in order to qualify for participation in this study. Subjects taking BOTH metformin and a sulfonylurea are not qualified for the trial.
  * Subjects must wash out from the following medications during the 7-day period prior to first dose, and must remain off these medications through discharge from period 4: metformin, sulfonylureas, statins, fat absorption blocking agents, bile acid sequestrants
  * All other prescription or non-prescription drugs, including vitamins, herbal and dietary supplements (including St John's Wort) are prohibited within 7 days or 5 half-lives (whichever is longer) prior to the first dose of study medication and through discharge from Period 4.
* Unwilling to abstain from

  * Caffeine-or xanthine-containing products for 24 hours prior to dosing until the final post-dose assessment at each treatment level
  * Use of illicit drugs
  * Alcohol for 24 hours prior to dosing until final post-dose assessment at each treatment level
  * Consumption of red wine, Seville oranges, grapefruit or grapefruit juice from 7 days prior to the first dose of study medication until collection of the final pharmacokinetic and pharmacokinetic blood samples
* History of sensitivity to any of the study medications, or components thereof or a history of drug or other allergy that, in the opinion of the physician responsible, contraindicates their participation. This includes sensitivity to heparin, if heparin will be used to maintain catheter patency.
* Where participation in the study would result in donation of blood in excess of 500 mL within a 56 day period.
* Subject is either an immediate family member of a participating investigator, study coordinator, employee of an investigator; or is a member of the staff conducting the study.

Ages: 18 Years to 60 Years | Sex: All | Healthy Volunteers: Yes
Age Groups: Adult
Enrollment: 36 (Actual)
Dates: Start 2007-11-16 (Actual); Primary Completion 2008-03-10 (Actual); Study Completion 2008-03-10 (Actual)

PRIMARY OUTCOMES:
adverse events: | each visit
clinical laboratory: | day -1, day 2 each period
electrocardiogram (ECG): | day 1 each period
vital signs assessments: | day -1, day 1 each period

SECONDARY OUTCOMES:
plasma drug concentrations: | Day 1 each dosing level
plasma blood sugar & other parameter concentrations: | Day 1 Period 4 following meal
Correlation between drug concentrations & blood sugar levels: | day 1 period 4

CONTACTS AND LOCATIONS:
Overall Officials: GSK Clinical Trials, Study Director — GlaxoSmithKline
Locations (1):
- GSK Investigational Site, Minneapolis, Minnesota, United States

IPD SHARING:
Plan to Share IPD: Yes
Patient-level data for this study will be made available through www.clinicalstudydatarequest.com following the timelines and process described on this site.

REFERENCES:
- See also: Researchers can use this site to request access to anonymised patient level data and/or supporting documents from clinical studies to conduct further research. — https://www.clinicalstudydatarequest.com
- See also: Results for study AXO110461 can be found on the GSK Clinical Study Register. — https://gsk-clinicalstudyregister.com/study/AXO110461?search=study&study_ids=AXO110461#rs
- Available data/document: Study Protocol: AXO110461 — https://www.clinicalstudydatarequest.com — For additional information about this study please refer to the GSK Clinical Study Register
- Available data/document: Annotated Case Report Form: AXO110461 — https://www.clinicalstudydatarequest.com — For additional information about this study please refer to the GSK Clinical Study Register
- Available data/document: Dataset Specification: AXO110461 — https://www.clinicalstudydatarequest.com — For additional information about this study please refer to the GSK Clinical Study Register
- Available data/document: Clinical Study Report: AXO110461 — https://www.clinicalstudydatarequest.com — For additional information about this study please refer to the GSK Clinical Study Register
- Available data/document: Statistical Analysis Plan: AXO110461 — https://www.clinicalstudydatarequest.com — For additional information about this study please refer to the GSK Clinical Study Register
- Available data/document: Individual Participant Data Set: AXO110461 — https://www.clinicalstudydatarequest.com — For additional information about this study please refer to the GSK Clinical Study Register
- Available data/document: Informed Consent Form: AXO110461 — https://www.clinicalstudydatarequest.com — For additional information about this study please refer to the GSK Clinical Study Register